CLINICAL TRIAL: NCT02029469
Title: Ascension® Humeral Resurfacing Arthroplasty Follow-Up Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated due to PI leaving the institution
Sponsor: Ascension Orthopedics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP- HRA-001
Record Dates: First submitted 2012-04-25; First posted 2014-01-08 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Shoulder Arthritis Osteoarthritis; Rheumatoid Arthritis Shoulder; Acquired Deformity of Head; Post-traumatic Arthrosis of Other Joints, Shoulder Region
Keywords: Humeral Resurfacing; Humeral Resurfacing Arthroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HRA Device (Experimental): Patients who will be treated with Ascension HRA device.
  Interventions: Device: Ascension HRA device

INTERVENTIONS:
Device: Ascension HRA device — Patients who are treated with the Ascension® HRA for resurfacing of humeral head.
  Other Names: Ascension Metal HRA device

SUMMARY:
It is a non-randomized, consecutive enrollment, 10-year follow-up study of patients who are treated with the Ascension® HRA. Its purpose is to measure and document the outcomes associated with implanting the Ascension HRA prosthesis. Patients will be periodically assessed to collect data related to safety and effectiveness endpoints at the following intervals: preoperative, surgery/immediate post-op, 3 months, 6 months, 1 year, 2 year, 5 year, and 10 years.

DETAILED DESCRIPTION:
At each assessment interval, information on complications and adverse events will be collected. In addition, shoulder joint range of motion will be collected, and implants will be evaluated radiographically to determine joint position and assess implant with regards to radiolucencies, subsidence and subluxation (migration). Patient satisfaction with regard to the effect of the implant on shoulder function, joint pain, and overall satisfaction will be assessed using a visual analog scale (VAS). Furthermore, if there are any implant revisions during the 10-year follow-up for any of the patients enrolled in the study, the implant and/or surrounding tissue will be harvested if possible and submitted for histopathological examination.

ELIGIBILITY:
Inclusion Criteria:

* The following patient will be included in the study - Patient who:

  * Is treated with the Ascension HRA;
  * Is disabled by either non-inflammatory or inflammatory arthritis (i.e. rheumatoid arthritis, osteoarthritis and avascular necrosis;
  * Has mild or moderate humeral head deformity and /or limited motion;
  * Has post-traumatic arthritis;
  * Has an intact or reparable rotator cuff;
  * Has the means and ability to return for all required study visits
  * Is willing to participate in the study;
  * Has signed an Informed Consent Form;
  * Is at least 18 years of age and skeletally mature at the time of surgery;
  * Is less than 75 years of age at the time of surgery

Exclusion Criteria:

The following patients will be excluded from the study - Patients who:

* Infection, sepsis, and osteomyelitis;
* Osteoporosis;
* Metabolic disorders which may impair bone formation;
* Osteomalacia;
* Rapid joint destruction, marked bone loss or bone resorption apparent on X-ray;
* Revision procedures where other devices or treatments have failed
* Refuses to be in the study; or does not have the means and ability to return for all required study visits;
* Currently participating in another clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2007-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
American Shoulder and Elbow Surgeon Score | Outcome data will be evaluated at 2 years
  The ASES score will be evaluated at 2 years and compared to baseline.

SECONDARY OUTCOMES:
Range of Motion | 2 years
  Shoulder range of motion will be measured compared to baseline.
VAS scale for pain | 2 years
  VAS score for pain will be evaluated at 2 years and compared to baseline.
AP and axillary radiographs | 2 years
  Radiographs will be evaluated at 2 years for subsidence, lucent lines and evidence of movement or pending failure.
Adverse events | 2 years and during entire trial
  AEs will be assessed at each study timepoint

CONTACTS AND LOCATIONS:
Overall Officials: Sam Hakki, M.D., Principal Investigator — Bay Pines VA Health Care System
Locations (1):
- Bay Pines VA Healthcare System, Bay Pines, Florida, United States